CLINICAL TRIAL: NCT06736002
Title: Effects of Mega-dose Vitamin D Pulse and Maintenance Therapy on Seizure Frequency, Fatigue, and Quality of Life: a Prospective Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chin-Wei Huang (Other)
Responsible Party: Sponsor-Investigator, Chin-Wei Huang, Professor, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-BR-113-028
Record Dates: First submitted 2024-11-28; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Epilepsy
Keywords: Mega-Vitamin D; Epilepsy; Fatigue; Quality of life
MeSH Terms: conditions — Epilepsy; Fatigue | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: RCT study with Mega-Vitamin D compare placebo Experimental group: Mega-Vitamin D 100.8 million IU for three months Control group: placebo for three months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental)
  Interventions: Other: Vitamin D; Other: Placebo
- Placebo (Placebo Comparator)
  Interventions: Other: Vitamin D; Other: Placebo

INTERVENTIONS:
Other: Vitamin D — Vitamin D
Other: Placebo — Placebo oral solution

SUMMARY:
We inform consent overall process of this trial study through face-to-face use of the IRB, clarify patient questions, and allow subjects to fully understand the trial study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 or above (inclusive)
* Diagnosed patients (refractory epilepsy refers to those who have used more than two drugs, and each drug has reached the When epileptic seizures cannot be well controlled at standard reasonable treatment doses, it is called refractory epilepsy)
* There is no imaging evidence of persistence or expansion of brain damage in the past three years
* Subjects or family members (caregivers) can comply with the trial plan and take vitamin D patients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
seizure frequency | three time points: before starting the medication, one month after starting the medication, and three months after starting the medication.
  The study aims to evaluate four major measurement indicators. First, the frequency of epileptic seizures will be assessed at three time points: before starting the medication, one month after starting the medication, and three months after starting the medication. This will allow for monitoring changes in seizure frequency and evaluating the effectiveness of the treatment over time.

SECONDARY OUTCOMES:
Quality of life | before starting the medication and again three months after treatment
  Second, quality of life will be assessed using the World Health Organization Quality of Life (WHOQOL-BREF) scale. Evaluations will be conducted before starting the medication and again three months after treatment, enabling a comparison of any improvements or changes in quality of life resulting from the medication.
fatigue | before starting the medication and three months after starting it.
  Third, fatigue will be evaluated using the Brief Fatigue Inventory (BFI). Measurements will take place before starting the medication and three months after starting it. This will provide insight into how the treatment impacts fatigue levels, which is important for understanding its overall effect on patient well-being.
Serum tests | three time points: before starting the medication, one month after starting it, and three months after starting it.
  Finally, serum levels of Vitamin D, Calcium (Ca), Phosphorus (P), and Parathyroid Hormone (PTH) will be measured at three time points: before starting the medication, one month after starting it, and three months after starting it. These tests will help to monitor any physiological changes or effects of the medication on key metabolic markers.

IPD SHARING:
Plan to Share IPD: No